CLINICAL TRIAL: NCT05337085
Title: To Compare Dexmedetomidine and Midazolam for Intra-op Sedation in TIVA in Children Undergoing Inguinal Hernia Repair
Brief Title: Comparison of Dexmedetomidine and Midazolam for Intra-op Sedation in TIVA in Children Undergoing Inguinal Hernia Repair
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Anab Farooqi, Dr. Anab Farooqi, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AFarooqi
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Inj. Dexmedetomidine (precidex) 200/mcg/2ml given to participants in infusion form for 10 mins of surgery and maintenance dose given till the end of surgery
  Interventions: Drug: Dexmedetomidine
- Midazolam (Active Comparator): Inj midazolam 0.5 mg/kg stat dose will be given to participants during surgery
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Inj dexmedetomidine and inj midazolam given to 2 groups of participants and sedative effects of both drugs will be observed during surgery
  Arms: Dexmedetomidine
Drug: Midazolam — Midazolam
  Arms: Midazolam

SUMMARY:
To compare dexmedetomidine and midazolam for intra-op sedation in TIVA in children undergoing inguinal hernia repair. The results of the study if found significant will guide the anesthetist in appropriate choice and dose of sedative drug with highest efficacy and minimum side effects to avoid post operative adverse effects associated with anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Male and female paediatric patients In age range neonates to 15 years
* Planned for elective inguinal hernia repair
* Patients with uncomplicated hernia With ASA class I or II

Exclusion Criteria:

* Patients undergoing emergency inguinal repair
* Patients with ASA class III,IV,V or VI
* Patients present with complicated hernia
* Patients with BMI above 40kg/m2
* Patients with any allergy to anesthesia
* Patients with coagulopathy
* Patients with narcotic/opioid addiction

Ages: 12 Months to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Level of sedation assessed through Ramsay Sedation Scale RSS | 6 months

IPD SHARING:
Plan to Share IPD: No